CLINICAL TRIAL: NCT06383364
Title: The Effect of a Medication Coordinator on the Quality of Patients Medication Treatment (MEDCOOR) - Randomized Controlled Trial
Brief Title: The Effect of a Medication Coordinator on the Quality of Patients Medication Treatment
Acronym: MEDCOOR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SHS-Pharm - 1 - 2024
Record Dates: First submitted 2024-03-18; First posted 2024-04-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Medication Review; Polypharmacy; Potentially Inappropriate Medication; Quality of Life; Medication Therapy Management
Keywords: Polypharmacy; Medication review; Patient care management; Empowerment; Potentially inappropriate medication list; Hospital to home transition; Medication quality; medication optimization; Treatment burden
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventions group (Active Comparator): The Medication Coordinator facilitates the medication reviews in close collaboration with the patients by applying concepts of motivational interview in combination with My Medication Plan
  Interventions: Behavioral: Medication Coordinator
- Control group (No Intervention): Usual treatment from a team consisting of hospital physicians, nurses, nurse assistants, and as needed occupational therapists, physiotherapist, and clinical dieticians. Medication reconciliation might be a part of the patients' usual care performed by physicians or pharmacologist present at the acute ward. Hospital physicians and/or nurses might perform patient counselling about medication treatment during hospitalization

INTERVENTIONS:
Behavioral: Medication Coordinator — The Medication Coordinator calls the patient app seven days after discharge in the transition of care from hospital to home
  Arms: Interventions group

SUMMARY:
To examine the effect of a Medication Coordinator, who facilitates medication reviews in close collaboration with patients using My Medication Plan to reduce the risk of post-hospital inappropriate medication usage.

DETAILED DESCRIPTION:
Patients' safety can be compromised in the transition of care between healthcare sectors. Optimal information flow across healthcare sectors and individualized medication treatment tailored to each patient is key to prevent adverse events and optimize patient treatment. Particularly, the inclusion of the general practitioner is important in this process; it could become a challenge to keep medication changes if this communication link is missing. The framework for complex intervention allows flexibility and adaption in meeting patients' needs by implementing tailored, possibly complex interventions in different healthcare settings. To examine the effect of a Medication Coordinator, who facilitates medication reviews in close collaboration with patients using My Medication Plan. The primary outcome is the proportion of potentially inappropriate medications. Secondary outcomes include patient-reported outcomes i.e., quality of life and medication burden. Additional outcomes include the patient's individual Medication Risk Score, if the patients are readmitted, and if the patients have contacted the staff at the hospital unit after the hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* all hospitalized patients, who are prescribed at least five medications specified in the Electronic Patient Journal (EPJ) used at ward

Exclusion Criteria:

* unable to communicate in Danish, cognitively impaired e.g. suffering from dementia or Alzheimer's, or cannot cooperate due to e.g. hallucination or aggressive behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in potentially inappropriate medication according to Potentially Inappropriate Medication List | Baseline and 6 months
  Evaluating the patients drug treatment to assess if a drug is a potentially inappropriate medication

SECONDARY OUTCOMES:
Evaluation of patients experiences quality of life with the EQ-5D and EQ-VAS. | Baseline and 3 months
  EQ-5D contains five questions regarding five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression each with five answer categories: no problems, slight problems, moderate problems, severe problems, and extreme problems. Permission for using the Danish EQ-5D version have been granted by EuroQol.
  The EQ-VAS is a vertical VAS with the patient reporting their perceived quality of life from 0-100 (60). The endpoints are labelled with "The worst health you can imagine" (0) and "The best health you can imagine" (100). This VAS is used to quantify the measure of health that reflects the patient's own perception.
Evaluation of patients experienced quality of life with visual analogue scale (VAS). | Baseline and 3 months
  The patients are to score their experienced VAS regarding quality of life with VAS.
  The VAS is a vertical VAS and ranges from zero (low quality of life) to 100 (the highest quality of life) by numbers. The endpoints are label with "The worst quality of life you can image" (0) and "The highest quality of life you can image" (100).
Evaluation of patients experienced treatment burden with the questionnaire Multimorbidity treatment burden questionnaire (MTBQ). | Baseline and 3 months
  The MTBQ is a validated tool to assess patients perceived treatment burden. Treatment burden is described as patients perception of the effort required to look after their health and the effect of this on their everyday life. A Danish version of the MTBQ has been validated and is applied upon permission.
  The MTBQ is a ten-item questionnaire with good content validity, high internal reliability, and good construct validity. The questions covers aspects of medication management self-monitoring, contact with healthcare professionals, obtaining information, implementing life-style changes, and relying on help. The answers are a five point Likert scale with the possibilities: "Not difficult" (0), "A little difficult" (1), "Quite difficult" (2), "Very difficult" (3), "Extremely difficult" (4), and "Does not apply" (0). The MTBQ scores are categorized into no burden (score 0), low burden (score < 10), medium burden (score 10-22), and high burden (score ≥ 22).
Evaluation of patients experienced medication burden with visual analogue scale (VAS). | Baseline and 3 months
  An additional VAS regarding treatment burden is added. The VAS is a vertical VAS and ranges from zero (no burden at all) to 100 (the highest burden imagined) by numbers. The endpoints are labelled with "The worst burden you can imagine" (0) and "The highest burden you can imagine" (100).
Patient readmission 30 days after hospital discharge | 30 days after the patient has been discharged from the hospital.
  Patient readmissions are evaluated 30 days after hospital discharge. As a "did" or "did not" and a time-to-event, with a restriction of 30 days. The readmissions are assessed through the electronic patient journal.
Patient contact to the ward 30 days after hospital discharge | 30 days after the patient has been discharged from the hospital.
  Patient contact to the ward are evaluated 30 days after hospital discharge. As a "did" or "did not" and a time-to-event, with the restriction of 30 days. And if possible to assess which question the patient had to the ward, if it was drug-related or more disease specific. The readmission are assessed through the electronic patient journal.

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schlunsen M, Graabaek T, Pedersen AK, Kampmann JD, Kjeldsen LJ. Study protocol: The effect of a Medication Coordinator on the quality of patients' medication treatment (MEDCOOR)-Randomized controlled trial. PLoS One. 2024 Nov 26;19(11):e0314023. doi: 10.1371/journal.pone.0314023. eCollection 2024. PMID 39591420